CLINICAL TRIAL: NCT00343395
Title: A Single-Center, Randomized, Double-Blind, Placebo-Controlled Clinical Trial of Combined Rosiglitazone/Metformin (Avandamet®) vs. Placebo on Serological Outcomes in Non-Diabetic Patients With Stable Coronary Syndromes
Brief Title: Rosiglitazone and Metformin: Outcomes Trial in Nondiabetic Patients With Stable Coronary Syndromes (Romance) Pilot Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: FDA concerns regarding Avandamet
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: J. Brent Muhlestein, MD, Intermountain Healthcare
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 128-013
Record Dates: First submitted 2006-06-21; First posted 2006-06-23 (Estimated); Last update posted 2011-03-17 (Estimated); Status verified 2011-03

CONDITIONS: Coronary Artery Disease
Keywords: rosiglitazone; metformin; hs-CRP; inflammation
MeSH Terms: conditions — Coronary Artery Disease; Inflammation | interventions — rosiglitazone-metformin combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Avandamet (Active Comparator): AVANDAMET 2/500 mg
  Interventions: Drug: AVANDAMET
- Placebo (Placebo Comparator)
  Interventions: Drug: AVANDAMET

INTERVENTIONS:
Drug: AVANDAMET — 2/500 mg

SUMMARY:
Nearly half of all Americans will die from cardiovascular disease caused by the build up of atherosclerotic plaque within coronary arteries. Most deaths in these patients arise from the development of acute coronary syndromes (ACS) such as myocardial infarction, unstable angina, or sudden death. ACS is characterized by coronary plaque erosion or rupture, which is triggered by endothelial changes, including inflammation, and thrombosis. Diabetes, with insulin resistance as a major component, has been shown to engender adverse metabolic events within the endothelial cell [1], including impaired endothelial function, augmented vasoconstriction, increased inflammation and thrombosis. Activation of the transcription factors nuclear factor KB (NF-KB) and activator protein 1 (AP-1) induces inflammatory gene expression, with liberation of leukocyte-attracting chemokines, increased production of inflammatory cytokines, and augmented expression of cellular adhesion molecules. These metabolic processes may therefore play a significant role in the development of ACS.The hypothesis is that rosiglitazone and metformin, or the combination of both may provide positive anti-atherogenic effect, even among patients without diabetes. This pilot study proposes to evaluate the effect of placebo vs. combined rosiglitazone/metformin (Avandamet®) on surrogate blood markers of atherosclerosis activity among non-diabetic and pre-diabetic patients with known stable coronary syndromes. This will provide further evidence justifying a large definitive outcomes-based clinical trial.

DETAILED DESCRIPTION:
This is a single-center, randomized, double-blind trial comparing combined rosiglitazone/metformin (Avandametä) to placebo in subjects with normal or intermediate fasting glucose (IFG) and stable coronary artery disease.Subjects meeting entry criteria will be randomized in a 1:1 ratio to receive either placebo or combined rosiglitazone/metformin (Avandametä) 4/1000 mg. Laboratory specimens including high sensitivity C-reactive protein (hs-CRP), glucose, HgbA1C, complete lipid profile, will be obtained after a 10 hour fast as specified by study visits. Subjects will return for repeat study visits at 2, 4, 6 and 8 months for repeat laboratory evaluations, including safety labs consisting of serum creatinine, liver enzymes, and a CBC. Additionally, subjects will have IL-6 and TNF-a measured for research purposes at baseline and subsequent follow-up visits. All subjects will be followed for a minimum of 8 months. This pilot study proposes to evaluate the effect of placebo, or combined rosiglitazone/metformin onsurrogate blood markers of atherosclerosis activity among non-diabetic and pre-diabetic patients with known stable coronary syndromes.

ELIGIBILITY:
Inclusion Criteria:

* The patient (male or non-pregnant female) must be > 18 years of age.
* The patient or legally authorized representative must sign a written informed consent, prior to the procedure, using a form that is approved by the local Institutional Review Board.
* Angiographically documented coronary artery disease defined as the presence of at least one 50% or greater stenosis of a major coronary artery.
* Stabilized post any prior ACS event (i.e., without ongoing ischemic rest pain, congestive heart failure, or malignant arrhythmias) for at least 3 months
* Fasting blood glucose 87-125 mg/dL

Exclusion Criteria:

* Age <18 years
* Known hypersensitivity to metformin or rosiglitazone
* Renal insufficiency defined as calculated creatinine clearance (CrCl) <40 mL/min using the following formula:

Men: CrCL (mL/min) = Weight (kg) x (140-age) 72 x serum creatinine (mg/dL) Women: 0.85 x the value calculated for men

* Pregnant and/or lactating women, and women of child bearing potential are excluded from this trial
* Co-morbidity such that the patient is not expected to survive >2 years
* Current therapy with rosiglitazone or metformin
* PCI within the previous six months (other than for the qualifying event)
* Prior CABG within the previous two months, scheduled CABG, or a decision to perform CABG made prior to enrollment
* Overt diabetes mellitus (FBG>126 or antidiabetic therapy)
* Any diagnosis of congestive heart failure
* Obstructive hepatobiliary disease or other significant hepatic disease (defined as the presence of at least one of the following: AST, ALT, GGT, total bilirubin, or alkaline phosphatase >3x upper limit normal, not related to MI
* Participation in any other clinical trials involving investigational or marketed products within 30 days prior to entry in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2006-06; Primary Completion 2007-11 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
To demonstrate the effect (change from baseline) of each study intervention on hs-C-reactive protein. | Study completion
To demonstrate the safety of the interventions on clinical outcomes (death, MI, cardiovascular hospitalizations) and serious drug-related adverse events. | Study completion

SECONDARY OUTCOMES:
To demonstrate the effect (change from baseline) of each study intervention on lipid levels | Study completion
To demonstrate the effect (change from baseline) of each study intervention on inflammatory marker levels other than hs-CRP | Study completion
To demonstrate the effect (change from baseline) of each study intervention on HgbA1C | Study completion
To demonstrate the effect (change from baseline) of each study intervention on fasting blood glucose | Study completion
Safety: Differences in adverse events between the two arms | Interim; completion of study

CONTACTS AND LOCATIONS:
Overall Officials: Joseph B Muhlestein, MD, Principal Investigator — Intermountain Healthcare, LDS Hospital
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States